CLINICAL TRIAL: NCT06162325
Title: The Efficacy and Safety of Venetoclax in Combination With Standard Induction and Consolidation Chemotherapy in Newly Diagnosed Young Acute Myeloid Leukemia
Brief Title: Venetoclax in Combination With Standard Induction and Consolidation Chemotherapy in Newly Diagnosed Young AML Patients
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: AML-VEN PLUS
Record Dates: First submitted 2023-12-01; First posted 2023-12-08 (Actual); Last update posted 2023-12-08 (Actual); Status verified 2023-12

CONDITIONS: Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational study is to to evaluate the efficacy and safety of Venetoclax in combination with DA60(daunorubicin 60 mg/m2/d for 3 days, and cytarabine 100 mg/m2 every 12 h for 7 days) induction and HD-AraC(cytarabine 3 g/m2 every 12 h for 3 days) consolidation, in young patients with newly diagnosed acute myeloid leukemia (AML).

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed, morphologically documented AML based on the World Health Organization (WHO) 2016 classification.
* Age ≥ 18 years and ≤ 59 years
* Have been treat with the "venetoclax in combination with standard induction and consolidation chemotherapy" therapy, and in follow-up.
* Be comprehensive of the research, and able to provide informed consent.

Exclusion Criteria:

* Diagnosis of acute promyelocytic leukemia (APL).
* Prior treatment for AML, except for: leukapheresis, hydroxyurea, and growth factor/cytokine.
* Unable to understand or participate.

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Newly diagnosed acute myeloid leukemia (AML) patients of the age 18 to 59 years old.
Sampling Method: Probability Sample
Enrollment: 45 (Estimated)
Dates: Start 2022-01-21 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Disease-free survival (DFS) | Assess up to 24 months.
  DFS is calculated from the date of remission (inclusive of CR and CRi) to the date of relapse, death from any cause, or last follow-up.

SECONDARY OUTCOMES:
Complete remission (CR) rate | On Day 21 (window Day 21 to Day 35), a bone marrow aspirate specimen will be collected for morphology and pathology.
  The rate of patient who get CR after induction therapy.
Rate of minimal residual disease (MRD) negativity | MRD will be tested after every cycle of therapy and during follow-up.
  Percentage of patients achieving CR with no evidence of MRD after induction therapy, 1 cycle of consolidation therapy, and 4 cycles of consolidation therapy. MRD negativity is defined as < 0.1% of CD45 expressing cells with the target immunophenotype, or as cycling threshold (Ct) ≥ 40 in ≥ 2 of 3 replicates by qPCR.
Overall survival (OS) | Assess up to 24 months.
  OS is defined as the duration from initiation of induction treatment to the date of death from any cause or last follow-up.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China